CLINICAL TRIAL: NCT05098366
Title: Utilization of Furosemide to Expedite Bladder Filling in Pediatric Females With Suspected Ovarian Torsion Awaiting Pelvic Ultrasound
Brief Title: Furosemide Use to Fill the Bladder of Pediatric Females Awaiting Pelvic Ultrasound
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, Candice Jersey, Pediatric Emergency Medicine Fellow, Connecticut Children's Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 21-008
Record Dates: First submitted 2021-08-05; First posted 2021-10-28 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Ovarian Torsion
Keywords: Pediatric; Point-of-care Ultrasound; Bladder volume
MeSH Terms: conditions — Ovarian Torsion | interventions — Furosemide; Saline Solution; Fluid Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Furosemide (Experimental): Participants will receive a 20mL/kg (max 1000mL) IV fluid bolus and a 0.1mg/kg (max 5mg) furosemide dose
  Interventions: Drug: Furosemide
- IV fluids (Placebo Comparator): Participants will receive a 20mL/kg (max 1000mL) IV fluid bolus and an IV fluid flush
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Furosemide — 0.1mg/kg (max 5mg) of IV furosemide
  Other Names: Lasix
  Arms: Furosemide
Drug: Normal saline — 20mL/kg (max 1000mL) normal saline bolus plus a normal saline flush
  Other Names: Intravenous fluids; IV fluids
  Arms: IV fluids

SUMMARY:
The purpose of this study is to investigate whether or not furosemide causes the bladder to fill faster than IV fluids alone so that a pelvic ultrasound exam can be performed.

DETAILED DESCRIPTION:
Trans-abdominal pelvic ultrasound is the standard imaging modality for diagnosis of ovarian torsion in the pediatric population, however this requires that the patient have a full bladder at the time of imaging. This study will investigate whether low dose furosemide in addition to IV fluid boluses may provide a fast, effective, and non-invasive means to fill the bladder of pediatric females awaiting pelvic US. The target population are females age 8 to 18 years seen in the emergency room at Connecticut Children's Medical Center who are undergoing a trans-abdominal pelvic ultrasound to assess for ovarian torsion. Enrolled patients will be randomized to the control (IVF bolus only) group vs. the intervention (IVF bolus + furosemide) group and will undergo point-of-care US (POCUS) and bladder scanner evaluation of the bladder every 30 minutes until the bladder is determined to be full.

ELIGIBILITY:
Inclusion Criteria:

1. Females age 8-18yrs seen in the ED at CCMC who are undergoing a trans-abdominal pelvic ultrasound to assess for ovarian torsion
2. Ability of patient (if 18yrs) or parent/legal guardian to sign a written informed consent

Exclusion Criteria:

1. History of renal, genitourinary, or pelvic anomalies

   a. Eg: Chronic kidney disease, anuria, vesicoureteral reflux, ureteral obstruction, urologic reconstructive surgery, suprapubic or pelvic surgery, indwelling urethral catheter, oophorectomy, bicornate uterus
2. Patients with multiple chronic illnesses or systemic neurologic abnormality

   a. Eg: Bronchopulmonary dysplasia, tracheostomy, gastrostomy tube dependence, cerebral palsy, severe developmental delay, mitochondrial disorder, congenital heart disease, cardiomyopathy, chronic kidney disease, diabetes
3. Patients with known pregnancy
4. Patients deemed to be critically ill

   a. Mental status changes, signs of end organ damage, hypotension
5. Contraindication to giving Furosemide

   a. Allergy to sulfonamide medications, severe dehydration, hypotension, underlying electrolyte abnormality, underlying renal disease
6. History of previous diuretic use within the past year
7. Patients who self-report their bladder as being full at the time of enrollment

Ages: 8 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2021-05-29 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The time from initiation of the intervention to the time that the bladder reaches large, ovoid shape on POCUS exam | Through study completion, about 3 hours
  Initiation of the intervention is defined as administration of furosemide vs. normal saline flush.

SECONDARY OUTCOMES:
The correlation between bladder volume as calculated on POCUS exam of a large, ovoid bladder and bladder volume as reported by bladder scanner | Through study completion, about 3 hours
  Measurements will be completed every 30 minutes through study completion
Number and nature of all reports of adverse events related to furosemide administration | From time of intervention until final disposition, about 6 hours
  Adverse events include signs of severe dehydration, allergic reaction, and electrolyte abnormality
The time from initiation of the intervention to the time of completion of successful radiology-performed pelvic US | About 3 hours
The time from initiation of intervention to the time of admission or discharge order placement | From time of intervention until final disposition, about 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Candice Jersey, D.O., Principal Investigator — Connecticut Children's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Prieto JM, Kling KM, Ignacio RC, Bickler SW, Fairbanks TJ, Saenz NC, Nicholson SI, Lazar DA. Premenarchal patients present differently: A twist on the typical patient presenting with ovarian torsion. J Pediatr Surg. 2019 Dec;54(12):2614-2616. doi: 10.1016/j.jpedsurg.2019.08.020. Epub 2019 Aug 30. PMID 31500875
- [Result] Guthrie BD, Adler MD, Powell EC. Incidence and trends of pediatric ovarian torsion hospitalizations in the United States, 2000-2006. Pediatrics. 2010 Mar;125(3):532-8. doi: 10.1542/peds.2009-1360. Epub 2010 Feb 1. PMID 20123766
- [Result] Childress KJ, Dietrich JE. Pediatric Ovarian Torsion. Surg Clin North Am. 2017 Feb;97(1):209-221. doi: 10.1016/j.suc.2016.08.008. PMID 27894428
- [Result] Naffaa L, Deshmukh T, Tumu S, Johnson C, Boyd KP, Meyers AB. Imaging of Acute Pelvic Pain in Girls: Ovarian Torsion and Beyond☆. Curr Probl Diagn Radiol. 2017 Jul-Aug;46(4):317-329. doi: 10.1067/j.cpradiol.2016.12.010. Epub 2016 Dec 21. PMID 28185689
- [Result] Karaman E, Beger B, Cetin O, Melek M, Karaman Y. Ovarian Torsion in the Normal Ovary: A Diagnostic Challenge in Postmenarchal Adolescent Girls in the Emergency Department. Med Sci Monit. 2017 Mar 15;23:1312-1316. doi: 10.12659/msm.902099. PMID 28296829
- [Result] Dessie A, Steele D, Liu AR, Amanullah S, Constantine E. Point-of-Care Ultrasound Assessment of Bladder Fullness for Female Patients Awaiting Radiology-Performed Transabdominal Pelvic Ultrasound in a Pediatric Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2018 Nov;72(5):571-580. doi: 10.1016/j.annemergmed.2018.04.010. Epub 2018 Jul 3. PMID 29980460
- [Result] Stranzinger E, Strouse PJ. Ultrasound of the pediatric female pelvis. Semin Ultrasound CT MR. 2008 Apr;29(2):98-113. doi: 10.1053/j.sult.2007.12.002. PMID 18450135
- [Result] Guerra LA, Keays MA, Purser MJ, Wang SY, Leonard MP. Pediatric cystogram: Are we considering age-adjusted bladder capacity? Can Urol Assoc J. 2018 Dec;12(12):378-381. doi: 10.5489/cuaj.5263. PMID 29940135
- [Result] Koff SA. Estimating bladder capacity in children. Urology. 1983 Mar;21(3):248. doi: 10.1016/0090-4295(83)90079-1. No abstract available. PMID 6836800
- [Result] Ross M, Selby S, Poonai N, Liu H, Minoosepehr S, Boag G, Eccles R, Thompson G. The Effect of a Full Bladder on Proportions of Diagnostic Ultrasound Studies in Children with Suspected Appendicitis. CJEM. 2016 Nov;18(6):414-419. doi: 10.1017/cem.2016.23. Epub 2016 Apr 4. PMID 27039941
- [Result] Shapira-Zaltsberg G, Fleming NA, Karwowska A, Trejo MEP, Guillot G, Miller E. Non-visualization of the ovaries on pediatric transabdominal ultrasound with a non-distended bladder: Can adnexal torsion be excluded? Pediatr Radiol. 2019 Sep;49(10):1313-1319. doi: 10.1007/s00247-019-04460-y. Epub 2019 Jul 9. PMID 31289908
- [Result] Ljungberg A, Segelsjo M, Dahlman P, Helenius M, Magnusson M, Magnusson A. Comparison of quality of urinary bladder filling in CT urography with different doses of furosemide in the work-up of patients with macroscopic hematuria. Radiography (Lond). 2021 Feb;27(1):136-141. doi: 10.1016/j.radi.2020.07.002. Epub 2020 Jul 26. PMID 32727709
- [Result] Helenius M, Segelsjo M, Dahlman P, et al. Comparison of four different preparation protocols to achieve bladder distension in patients with gross haematuria undergoing CT urography. Radiography 2012;18:206-11.
- [Result] Van Der Molen AJ, Cowan NC, Mueller-Lisse UG, Nolte-Ernsting CC, Takahashi S, Cohan RH; CT Urography Working Group of the European Society of Urogenital Radiology (ESUR). CT urography: definition, indications and techniques. A guideline for clinical practice. Eur Radiol. 2008 Jan;18(1):4-17. doi: 10.1007/s00330-007-0792-x. Epub 2007 Nov 1. PMID 17973110
- [Result] Eades SK, Christensen ML. The clinical pharmacology of loop diuretics in the pediatric patient. Pediatr Nephrol. 1998 Sep;12(7):603-16. doi: 10.1007/s004670050514. PMID 9761364
- [Result] Oh SW, Han SY. Loop Diuretics in Clinical Practice. Electrolyte Blood Press. 2015 Jun;13(1):17-21. doi: 10.5049/EBP.2015.13.1.17. Epub 2015 Jun 30. PMID 26240596